CLINICAL TRIAL: NCT05087004
Title: Planned Parenthood Great Northwest, Hawai'i, Alaska, Indiana, Kentucky Teen Council Program Study
Brief Title: Planned Parenthood Teen Council Program Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philliber Research & Evaluation (Other)
Responsible Party: Principal Investigator, Sally Brown, Senior Researh Associate, Philliber Research & Evaluation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Philliberresearch
Record Dates: First submitted 2021-09-30; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Adolescent Problem Behavior
Keywords: Adolescent pregnancy prevention; Youth development

STUDY DESIGN:
Intervention Model Description: Participating Planned Parenthood affiliates recruited teens to their Teen Council program each study year during the spring and summer months. Interested teens completed an application and, if after review they were deemed by the program to be good candidates, they were interviewed. Active consent was obtained from the parents or guardians of all eligible youth and teen assent was also collected. Twice as many qualified applicants as spots on each Teen Council were accepted and their names were submitted to Philliber for random assignment to the program or survey-only groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teen Council Pogram (Experimental): Teens assigned to the intervention group received a 1-year long Teen Council Program.
  Interventions: Behavioral: Teen Council
- Control Group (No Intervention): Teens assigned to the control group did not receive any intervention.

INTERVENTIONS:
Behavioral: Teen Council — Youth randomly selected for Teen Council attended weekly meetings for an entire school year to receive training on specific topics. In turn, they provided educational presentations to the community, which required that they miss school (about one day per month). The presentations Teen Council members offered in middle and high schools were most commonly on birth control methods; relationships; reproductive anatomy and physiology; sexual diversity; STDs/STIs; sexual consent; HIV/AIDS; and abstinence.
  Arms: Teen Council Pogram

SUMMARY:
This is a randomized controlled trial (RCT) evaluation of the Teen Council program that was tested with high school students (grades 10-12) to assess whether it results in a reduction of teen pregnancy among other outcomes.

DETAILED DESCRIPTION:
Over the course of five years, we expected to have approximately 800 teens (400 program and 400 control) in the study. Teens were randomly selected for the program (Teen Council) and control (no program) conditions.

Teens in both groups were surveyed in the late summer/early fall of their enrollment year and each spring thereafter. Participation in the evaluation by control teens and unenrolled program teens was recognized with a small stipend.

The pre-survey was administered during the summer retreat for incoming Teen Council members. The same survey was administered by Philliber staff for the control youth via online, telephone, or mailed surveys during the late summer/fall. The post-surveys were administered at the end of the school year. Again, the survey was administered by program facilitators for the Teen Council program group. Philliber administered the post survey for the control group providing the same options for completion (online, telephone, or mail).

To facilitate follow-up, complete contact information was collected at baseline. This included the telephone numbers, physical addresses, and email addresses of the student and telephone numbers of their parents/guardians. Also requested was contact information for two relatives or adult friends who would likely know how to contact the teen. Parents were asked on the consent form to provide permission to receive change of school information in the event that their teen transferred to a new school. Philliber reached out to unenrolled Teen Council members and control group teens by telephone, email, text messaging, and/or U.S. Mail for survey administration (via telephone, online, or hard copy).

ELIGIBILITY:
Inclusion Criteria:

Applicants had to be:

1. entering 10th, 11th, or 12th grades;
2. able to attend an annual mandatory overnight retreat;
3. interested in providing accurate sexual health information to peers;
4. able to commit to weekly meetings;
5. able to miss school occasionally for presentations (one day per month);
6. responsible for budgeting their time and keeping up with their academic work.

Exclusion Criteria:

Any interested participant who did not meet all of the inclusion criteria:

1. was not entering 10th, 11th, or 12th grades;
2. was not able to attend an annual mandatory overnight retreat;
3. was not interested in providing accurate sexual health information to peers;
4. was not able to commit to weekly meetings;
5. was not able to miss school occasionally for presentations (one day per month); (6) was not responsible for budgeting their time and keeping up with their academic work.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 810 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
Ever had sex | Prior to program participation (baseline)
  Study participants were asked, "Have you ever had sexual intercourse?" Sexual intercourse was defined as any oral, anal, or penis-in-vagina sex. Item response choices were Yes/No.
Ever had sex | 1 year
  Study participants were asked, "Have you ever had sexual intercourse?" Sexual intercourse was defined as any oral, anal, or penis-in-vagina sex. Item response choices were Yes/No.
Contraceptive use at last intercourse | Prior to program participation (baseline)
  Study participants were asked, "The last time you had sexual intercourse, which methods did you or your partner use to prevent pregnancy?" Item response options included: I have never had penis-in-vagina sexual intercourse; no method was used to prevent pregnancy; birth control pills; condoms; Depo-Provera (or any injectable birth control), Nuva Ring (or any birth control ring), Implanon (or any implant), birth control patch, or any IUD; withdrawal; some other method; and not sure. These responses were recoded to Yes/No.
Contraceptive use at last intercourse | 1 year
  Study participants were asked, "The last time you had sexual intercourse, which methods did you or your partner use to prevent pregnancy?" Item response options included: I have never had penis-in-vagina sexual intercourse; no method was used to prevent pregnancy; birth control pills; condoms; Depo-Provera (or any injectable birth control), Nuva Ring (or any birth control ring), Implanon (or any implant), birth control patch, or any IUD; withdrawal; some other method; and not sure. These responses were recoded to Yes/No.
Changes to contraceptive method in last year | Prior to program participation (baseline)
  Study participants were asked, "During the last year, have you made any changes in the use of protection from sexually-transmitted infections (STIs) or pregnancy? Item response categories included: I have never had sexual intercourse; I haven't had sexual intercourse in the past 12 months; no; yes. If response was yes, study participants were asked to identify their previous contraceptive method and their current contraceptive method. Contraceptive methods were coded as reliable or not reliable.
Changes to contraceptive method in last year | 1 year
  Study participants were asked, "During the last year, have you made any changes in the use of protection from sexually-transmitted infections (STIs) or pregnancy? Item response categories included: I have never had sexual intercourse; I haven't had sexual intercourse in the past 12 months; no; yes. If response was yes, study participants were asked to identify their previous contraceptive method and their current contraceptive method. Contraceptive methods were coded as reliable or not reliable.
Ever visited doctor/clinic for birth control, exam, or STI | Prior to program participation (baseline)
  Study participants were asked, "j. Have you ever been to a doctor or to a clinic to get birth control, to have a pelvic exam, a testicular exam or to get a check up for sexually transmitted infections?" Item responses were Yes/No.
Ever visited doctor/clinic for birth control, exam, or STI | 1 year
  Study participants were asked, "j. Have you ever been to a doctor or to a clinic to get birth control, to have a pelvic exam, a testicular exam or to get a check up for sexually transmitted infections?" Item responses were Yes/No.

SECONDARY OUTCOMES:
Comfort with own sexuality scale | Prior to program participation (baseline)
  Seven-items that measured such things as comfort talking with a date about sex or birth control and having a good understanding of one's own sexual feelings and reactions (alpha = 0.7545). Each item was rated on a scale of 1 to 4, with the most desirable response being 4.
Comfort with own sexuality scale | 1 year
  Seven-items that measured such things as comfort talking with a date about sex or birth control and having a good understanding of one's own sexual feelings and reactions (alpha = 0.7545). Each item was rated on a scale of 1 to 4, with the most desirable response being 4.
Confidence in peer education skills scale | Prior to program participation (baseline)
  Eight-items, on a scale of 1 to 4, that measured confidence in accessing current information about sexually transmitted diseases and infections or explaining proper condom usage to peers (alpha = 0.7525).
Confidence in peer education skills scale | 1 year
  Eight-items, on a scale of 1 to 4, that measured confidence in accessing current information about sexually transmitted diseases and infections or explaining proper condom usage to peers (alpha = 0.7525).
Civic action scale | Prior to program participation (baseline)
  Six-item scale adapted from Flanagan et al. to measure ability to be actively engaged citizens (alpha = 0.6789). The scale, rated on a scale of 1 to 4, measured such things as the strength of their belief that they can make a difference in their communities and confidence that they can express their views in front of a group.
Civic action scale | 1 year
  Six-item scale adapted from Flanagan et al. to measure ability to be actively engaged citizens (alpha = 0.6789). The scale, rated on a scale of 1 to 4, measured such things as the strength of their belief that they can make a difference in their communities and confidence that they can express their views in front of a group.
Perspective taking scale | Prior to program participation (baseline)
  Seven-item sub-scale from the Interpersonal Reactivity Index measuring the ability of youth to be empathetic and understand the perspective of others (alpha = 0.7158). This 5-point subscale included items to measure attempts to understand their friends by imagining how things look from their perspective and trying to look at both sides of every question. The scale language was adapted to be more gender neutral, with permission of the author.
Perspective taking scale | 1 year
  Seven-item sub-scale from the Interpersonal Reactivity Index measuring the ability of youth to be empathetic and understand the perspective of others (alpha = 0.7158). This 5-point subscale included items to measure attempts to understand their friends by imagining how things look from their perspective and trying to look at both sides of every question. The scale language was adapted to be more gender neutral, with permission of the author.
Communication with parents | Prior to program participation (baseline)
  Two items about teen comfort talking with parents about sex and birth control, rated 1 to 4, with 4 indicating the highest level of comfort. These two items were examined individually. A third item measured whether youth had conversations with parents about sexuality or birth control in the past year (yes/no). A final item had teens report the number of such conversations in five unequal categories (0,1-5, 6-10, 11-15, and more than 15), then dichotomized to 10 or fewer conversations (0) and more than ten conversations (1).
Communication with parents | 1 year
  Two items about teen comfort talking with parents about sex and birth control, rated 1 to 4, with 4 indicating the highest level of comfort. These two items were examined individually. A third item measured whether youth had conversations with parents about sexuality or birth control in the past year (yes/no). A final item had teens report the number of such conversations in five unequal categories (0,1-5, 6-10, 11-15, and more than 15), then dichotomized to 10 or fewer conversations (0) and more than ten conversations (1).

IPD SHARING:
Plan to Share IPD: No
Full study report is available upon request.